CLINICAL TRIAL: NCT02300766
Title: Nordic Study of the Cerebellar Mutism Syndrome in Children With Brain Tumours of the Posterior Fossa
Brief Title: Cerebellar Mutism Syndrome Study
Status: Recruiting | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Odense University Hospital (Other); Aarhus University Hospital (Other); Aalborg University Hospital (Other); Technical University of Denmark (Other); Karolinska University Hospital (Other); Skane University Hospital (Other); University Hospital, Linkoeping (Other); Uppsala University Hospital (Other); Sahlgrenska University Hospital (Other); University Hospital, Umeå (Other); Oslo University Hospital (Other); Trondheim University Hospital (Other); Haukeland University Hospital (Other); University Hospital of North Norway (Other); Helsinki University Central Hospital (Other); Tampere University Hospital (Other); Kuopio University Hospital (Other); Turku University Hospital (Other Government); Oulu University Hospital (Other); Radboud University Medical Center (Other); Liverpool University Hospitals NHS Foundation Trust (Other Government); Great Ormond Street Hospital for Children NHS Foundation Trust (Other); Nottingham University Hospitals NHS Trust (Other); University Hospital Birmingham (Other); University Hospitals Bristol and Weston NHS Foundation Trust (Other); Royal Infirmary of Edinburgh (Other); South Glasgow University Hospitals NHS Trust (Other); University Hospital Tuebingen (Other); Medical University of Vienna (Other); Ospedale Pediatrico Bambin Gesù (Other); Motol University Hospital (Other); University of Leipzig Medical Center (Unknown); Universitaire Ziekenhuizen KU Leuven (Other); Queen Fabiola Children's University Hospital (Other); Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other); University Hospital, Ghent (Other); Hospital De La Citadelle (Unknown); CHC MontLégia (Unknown); University Hospital, Antwerp (Other); Hospital Sant Joan de Deu (Other); Vienna University Hospital, Austria (Unknown)
Responsible Party: Principal Investigator, René Mathiasen, MD, PhD student, Rigshospitalet, Denmark
Other Study IDs: H-6-2014-002
Record Dates: First submitted 2014-11-21; First posted 2014-11-25 (Estimated); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Infratentorial Neoplasms; Mutism
Keywords: Cerebellar Mutism Syndrome; Posterior Fossa Tumor; Pediatric cancer; Neurosurgical techniques
MeSH Terms: conditions — Infratentorial Neoplasms; Mutism; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — A blood sample from each patient will be collected in order to make SNP analyses on the DNA to explore the role of genomic variants on the development, severity and recovery from the CMS.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Posterior fossa tumor patients: Children (0-18 years) with a tumour in the posterior fossa (cerebellum/4th ventricle/brainstem ) requiring surgery or open biopsy at one of the participating centres.

SUMMARY:
The purpose of this study is to determine why up to 25% of the pediatric patients who have surgery for a tumor in the posterior fossa develops the Cerebellar Mutism Syndrome (CMS). Furthermore the purpose is to explore the clinical course and the best treatment of the syndrome.

DETAILED DESCRIPTION:
Background:

Cancer accounts for 22 % of all deaths among children in Europe and is thus the leading non-traumatic pediatric cause of death. Central nervous system (CNS) tumours constitute 25% of all childhood cancers, and the majority of these are located in the posterior fossa. One of the most troublesome late effects after neurosurgery for such a tumour is the cerebellar mutism syndrome which is seen in up to 25% of the patients. It is characterized by mutism, hypotonia, ataxia and irritability. The exact aetiology, risk factors, clinical course and treatment have yet to be identified. The aim of this study is to accomplish that.

Method:

This is an observational prospective multicentre study that will include a minimum of 500 paediatric patients with posterior fossa CNS tumours from the Nordic countries. Additional countries might be added later once the study is running. The study has started in fall 2014 in 20 centres from 5 Nordic countries. Prior to this a pilot study was performed on 43 Danish adult patients to validate and fine-tune registration procedure. All patients will be treated according to local standards, but clinical data will be collected and imaging will be reviewed centrally.

To calculate the participation rate the annual number of included patients from each country will be compared to the number of registered patients in the cancer registers of the respective country and year.

A blood sample for genetic analysis will be collected from all patients. The patients' neurology and speech functions will be examined both pre-operatively and repeatedly post-operatively, including recording of standardised speech samples. All data will be collected trough a, for the purpose developed, online database.

Registration of data

The following data will be registered at the following 5 time points:

1. Preoperatively Hospital and country, and patient related variables (date of birth, handedness, bilingualism, sex and date of diagnosis). Medical history (Previous neurological/neuropsychological/ psychiatric problems, comorbidities, previous operations or other treatment for the tumour, previous regular use of any kind of medication). Preoperative neurological status will be examined and a language and speech test will be performed and recorded. If the patient is younger than 2 years a bedside assessment of the speech will be performed instead of a test. A blood sample for genetic analysis will be drawn together with the standard blood samples. Alternatively this can be done at any time during follow-up.
2. Postoperatively within 72 hours of surgery Operation related variables (date, duration and course of operation, surgical position, surgical approach, and tumour removal method), complications, technology employed, preoperative hydrocephalus and estimated completeness of tumour resection.
3. Postoperatively within 1-4 weeks from surgery Approximately 1-2 weeks post-op: Postoperative language and speech status and for those older than 2 years, a recording of a speech sample. Neurological examination. Glucocorticoid administration pre-, intra- or postoperatively plus other medications used to treat the CMS postoperatively and their effects. Kind(s) of imaging performed on the tumour pre- and postoperatively. Approximately 4 weeks post-op: Development and treatment of postoperative intracranial haematoma and hydrocephalus, leakage of cerebrospinal fluid and need for ventilator.
4. Postoperatively at about 2 months from surgery Postoperative development of CMS, detailed survey of the status of CMS in those affected including recording of speech sample and neurological examination. Medications used to treat the CMS since last registration and their effects.
5. Postoperatively at about 12 months from surgery Language and neurological status including a speech sample for those older than 2 years. Medications used to treat the CMS since last registration and their effects. Other anti-cancer treatment given (chemotherapy and/or radiotherapy). Results from the pathology department regarding the kind of tumour histology and genetics. Registration of whether neuropsychological assessment(s) have been performed. Kind(s) of imaging performed on the tumour since 1st follow-up. Copies of the MRIs and descriptions performed pre-op, right after the operation and approximately. 12 months post-op are obtained.

All registered data will be examined by a third party who will check for missing data or misentries in order to ensure a high quality of the data. In case of missing data or misentries the third party will contact the person who made the registration.

The database is administered by the children's cancer epidemiology group (CCEG) at Karolinska Hospital in Stockholm, which is also responsible for the Swedish children's brain tumour registry and the leukaemia database for the Nordic Society of Pediatric Hematology and Oncology (NOPHO)

Other courses:

In case of acute surgery, coma etc. information about the study and the offer to participate can be given within 7 days from the operation. In these cases preoperative data about the patient can be obtained from the patient's medical record and/or from the parents, but a preoperative speech sample cannot be performed. These patients will not be included in the analysis of whether and how preoperative speech and language status affects the risk of developing CMS, but will be included in all the other study analyses. Speech samples will be performed postoperatively in exactly the same manner as in patients that were included before operation to able to monitor the patient's speech postoperatively and register signs of the CMS.

Should the patient have posterior fossa tumour surgery performed again during the 12 months follow-up period, the patient will re-start the follow-up programme from that date. A separate pre-op and all the post-op registrations will be performed again, and used in the analysis of risk of first versus second or further surgery. New genetic blood samples will not be necessary in these cases. Should the patient have posterior fossa tumour surgery performed after the last 12 months follow-up, the patient will be offered to participate in the study again and a new consent will have to be obtained. New genetic blood samples will not be necessary in these cases.

If the patient leaves the study for any reason before the follow-up 12 months post-op, a separate form will be filled out explaining why the patient left.

If the patient turns 18 while included in the study, a new consent to participate will have to be given by the patient him- /herself.

Blood samples and analyses:

As soon as a patient has been registered, the study centre will request a 2 ml anticoagulated blood sample for genetic profiling (Single-Nucleotide Polymorphism (SNP) analysis).

The investigators will use a newly developed single nucleotide polymorphism (SNP) sequencing strategy that allows cost-effective mapping of 25-30.000 genetic polymorphisms within biological domains that could potentially be linked to the development of CMS (e.g. inflammation, vascularization, blood-brain-barrier markers, and apolipoprotein E and other lipoprotein pathway genes). The genetic data will be linked to the clinical data to identify genetic variants associated with the risk of CMS or the course of CMS. Specifically the investigators will map all SNPs in all genes that are known or are likely to be linked to these pathways, including mRNA binding sites and first order protein-protein interactions. Rather than expecting large effects of single SNPs, the strategy of this approach is to use front-line bioinformatics and pathway analyses to explore the additive effect of numerous SNPs involved in the same biological pathway. This will identify high-impact pathways, although with individual low-impact SNPs. The results obtained could guide future therapeutic approaches to CMS.

If the custodial parents do not consent to their child contributing a blood sample to the study, the child may still participate in the study, albeit not in the part involving genetic analysis. The samples as well as the rest of the study data will be protected under the Act on Processing of Personal Data and the Act on the Health Act.

All MRIs are analyzed by neuroradiologists with respect to tumour resection and neuroradiographic signs associated with CMS.

All speech recording are analyzed by speech therapists with respect to signs associated with CMS. The results of neuropsychological tests that may have been performed routinely will be separately obtained and analyzed.

Power calculations:

For the surgical hypothesis, assuming that 35% of patients are operated with an approach that has a lower risk of CMS (assumed to be 10%) and the remaining 65% of patients are operated using other approaches that carries a 20% risk of CMS, the investigators will with 80% power be able to identify a difference at a 5% significance level if the investigators include a total of 450 patients.

For the genetic analysis, several pathways and SNP-profiles will be explored with appropriate adjustments for multiple comparisons. Multiple SNPs will due to randomness be found to be related with the risk of CMS. Their true biological significance will subsequently be validated through internal validation, as the investigators will explore if other SNPs in the same biological pathway, e.g. SNPs in the same genes but not the same haplotype or SNPs that affect coding or regulatory regions in the identified risk-related genes are more significantly associated with risk of CMS than randomly selected SNPs. Furthermore, the genes/SNPs will be explored by bioinformatic predictions of the impact of the SNPs on protein-folding, binding affinity etc. Once such high-risk SNPs/genes/pathways have been identified and published, the investigators will attempt to have them confirmed in independent patient cohorts from Europe or the US. Based on a projected overall risk of CMS of 20%, a frequency of a specific SNP (or SNP-profile) of 30%, and a projected doubled risk of CMS in the group that harbour the SNP (or SNP-profile), the investigators will with 90% power be able to identify such a genetic predisposition at a 5% significance level, if a total of 343 patients are included in the study. Thus, the study has sufficient power.

To analyze the effect of the above mentioned variables (surgical method, administration of corticosteroid, handedness etc.) on the risk of developing CMS the investigators will perform univariate and multivariate regression analyses as well as standard descriptive analyses. These analyses will be performed using R.

Discussion:

The study will be the largest prospective multicenter study on cerebellar mutism syndrome to date, and the first one of its kind to systematically gather detailed information about 1) the surgical approaches least likely to cause the syndrome, 2) how the syndrome is best treated, 3) the role of genetics and 4) differences in incidence and clinical course of the syndrome for different patients.

The ultimate aim of the study is to reduce the incidence and improve the treatment of cerebellar mutism syndrome and lead to harmonization of the treatment of CNS tumour patients across the Nordic countries.

ELIGIBILITY:
Inclusion Criteria:

* Age < 18 years at the date of first imaging showing this tumour
* Tumour in the cerebellum/4th ventricle/brainstem with intention to treat with surgical resection or open biopsy. Second and further surgeries are also included.
* Informed consent from custodial parent(s)

Exclusion Criteria:

* None

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All children (0-18 years) with a tumour in the posterior fossa (cerebellum/4th ventricle/brainstem ) requiring surgery or open biopsy at one of the participating centres.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2014-10; Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Development and progress of Cerebellar Mutism Syndrome | 1 year after surgery
  The development of CMS is determined by a survey developed Robertson et al. The correlation between the risk of developing CMS and different neurosurgical techniques, genomic variants, treatments, tumor types, comorbidities, neuroradiologic findings, handedness and preoperative language status will be explored.

SECONDARY OUTCOMES:
Development and progress of reduced speech output | 1 year after surgery
  Speech production that is severely reduced and limited to single words or short sentences which can only be elicited after vigorous stimulation

CONTACTS AND LOCATIONS:
Overall Officials: Kjeld Schmiegelow, MD, Dr. med, Study Chair — Rigshospitalet, Denmark; Marianne Juhler, MD, Dr. med, Principal Investigator — Rigshospitalet, Denmark; Karsten Nysom, MD, Study Chair — Rigshospitalet, Denmark
Locations (30):
- Medical University of Vienna, Vienna, Austria
- University Hospital Leuven, Leuven, Belgium
- Motol University Hospital, Prague, Czechia
- Denmark (4):
  - Aalborg University Hospital, Aalborg
  - Aarhus University Hospital, Aarhus
  - Rigshospitalet, Copenhagen
  - Odense University Hospital, Odense
- Finland (5):
  - Helsinki University Central Hospital, Helsinki
  - Kuopio University Hospital, Kuopio
  - Oulu University Hospital, Oulu
  - Tampere University Hospital, Tampere
  - Turku University Hospital, Turku
- University of Leipzig Medical Center, Leipzig, Germany
- Semmelweis University, 2nd Dept of Pediatrics, Budapest, Hungary
- Ospedale Pediatrico Bambino Gesù, Rome, Italy
- Hospital of Lithuanian University of Health Sciences Kauno klinikos, Kaunas, Lithuania
- Netherlands (3):
  - Radboud University Nijmegen Medical Centre, Nijmegen, Gelderland
  - UMC Groningen, Groningen
  - UMC Utrecht, Utrecht
- Norway (4):
  - Haukeland University Hospital, Bergen
  - Oslo University Hospital, Oslo
  - University Hospital of North Norway, Tromsø
  - St. Olav's Hospital, Trondheim
- Sweden (6):
  - Sahlgrenska University Hospital, Gothenburg
  - Linköping University Hospital, Linköping
  - Skåne University Hospital, Skåne
  - Karolinska University Hospital, Stockholm
  - University Hospital of Umeå, Umeå
  - Uppsala University Hospital, Uppsala
- Alder Hey Childrens NHS Foundation Trust, Liverpool, United Kingdom

REFERENCES:
- [Derived] Laustsen AF, Fric R, Gronbaek JK, Benes V, Lopez VS, Nestler U, Carai A, Solanki G, Avula S, Malluci C, Nilsson P, Nyman P, Hjort MA, Brandsma R, Hoving E, Bua A, Taborska J, Mudra K, Balazs M, Rutkaiskiene G, Rocka S, Lemiere J, Wilhelmy F, Dorfer C, Sehested A, Juhler M, Mathiasen R. Preoperative hydrocephalus and the risk of postoperative speech impairment following posterior fossa tumour surgery in children: results from a prospective, multinational cohort study. Childs Nerv Syst. 2026 Feb 4;42(1):60. doi: 10.1007/s00381-026-07132-z. PMID 41639295
- [Derived] Laustsen AF, Gronbaek JK, Fric R, Avula S, Mallucci C, Nilsson P, Nyman P, Hauser P, Mudra K, Kiudeliene R, Rocka S, Hjort MA, Brandsma R, Hoving E, Carai A, Benes V, Taborska J, Dorfer C, Jacobs S, Pavon-Mengual M, Skjoth-Rasmussen J, Schmiegelow K, Sehested A, Mathiasen R, Juhler M. Postoperative speech impairment and cranial nerve deficits in children undergoing posterior fossa tumor surgery with intraoperative MRI - a prospective multinational study. Acta Neurochir (Wien). 2025 Sep 22;167(1):252. doi: 10.1007/s00701-025-06669-3. PMID 40982141
- [Derived] Sarup R, Laustsen AF, Sorensen MK, Mallucci C, Pizer B, Aquilina K, Molinari E, Hjort MA, Fric R, Nyman P, Sabel M, Nilsson P, Matukevicius A, Hauser P, Mudra K, Carai A, Zipfel J, Hoving E, van Baarsen K, IIIrd VB, Peyrl A, Nysom K, Sehested AM, Schmiegelow K, Juhler M, Gronbaek JK, Mathiesen R. Glucocorticoid use in paediatric posterior fossa tumour surgery and the occurrence of postoperative speech impairment. Childs Nerv Syst. 2025 Jul 11;41(1):231. doi: 10.1007/s00381-025-06850-0. PMID 40643729
- [Derived] Laustsen AF, Avula S, Gronbaek J, Pizer B, Nyman P, Nilsson P, Fric R, Hjort MA, Benes V, Hauser P, Palmafy B, Rutkauskiene G, Wilhelmy F, Brandsma R, Sehested A, Mathiasen R, Juhler M. Tumour volume as a predictor of postoperative speech impairment in children undergoing resection of posterior fossa tumours: a prospective, multicentre study. Acta Neurochir (Wien). 2025 Apr 3;167(1):97. doi: 10.1007/s00701-025-06459-x. PMID 40178678
- [Derived] Wibroe M, Cappelen J, Castor C, Clausen N, Grillner P, Gudrunardottir T, Gupta R, Gustavsson B, Heyman M, Holm S, Karppinen A, Klausen C, Lonnqvist T, Mathiasen R, Nilsson P, Nysom K, Persson K, Rask O, Schmiegelow K, Sehested A, Thomassen H, Tonning-Olsson I, Zetterqvist B, Juhler M. Cerebellar mutism syndrome in children with brain tumours of the posterior fossa. BMC Cancer. 2017 Jun 21;17(1):439. doi: 10.1186/s12885-017-3416-0. PMID 28637445